CLINICAL TRIAL: NCT00704405
Title: A Phase II Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of 4 Different Regimens of MK-7009 When Administered Concomitantly With Pegylated Interferon and Ribavirin in Treatment-Experienced Patients With Chronic Genotype 1 Hepatitis C Virus Infection
Brief Title: Safety and Efficacy of Vaniprevir (MK-7009) With Pegylated Interferon (Peg-IFN) and Ribavirin (RBV) in Treatment-Experienced Hepatitis C Virus (HCV) Participants (MK-7009-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-009; 2007_659 (Other: Merck Registration Number)
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — vaniprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 24-wk Vaniprevir 600 mg + Peg-IFN/RBV (Experimental): Vaniprevir 600 mg (total daily dose) and RBV (1000 mg or 1200 mg total daily dose based on body weight) twice daily (b.i.d.) and Peg-IFN 180 mcg injection once weekly for 24 weeks.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (Peg-IFN); Drug: Ribavirin (RBV)
- 24-wk Vaniprevir 600 mg + 24-wk PBO + Peg-IFN/RBV (Experimental): Vaniprevir 600 mg (total daily dose) and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for 24 weeks, followed by PBO and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for an additional 24 weeks.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (Peg-IFN); Drug: Ribavirin (RBV); Drug: Placebo (PBO)
- 48-wk Vaniprevir 300 mg + Peg-IFN/RBV (Experimental): Vaniprevir 300 mg (total daily dose, taken once daily [q.d.]) and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for 48 weeks.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (Peg-IFN); Drug: Ribavirin (RBV)
- 48-wk Vaniprevir 600 mg + Peg-IFN/RBV (Experimental): Vaniprevir 600 mg and RBV (1000 mg or 1200 mg based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for 48 weeks.
  Interventions: Drug: Vaniprevir; Drug: Pegylated Interferon (Peg-IFN); Drug: Ribavirin (RBV)
- 48-wk PBO + Peg-IFN/RBV (Placebo Comparator): PBO and RBV (1000 mg or 1200 mg based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for 48 weeks.
  Interventions: Drug: Pegylated Interferon (Peg-IFN); Drug: Ribavirin (RBV); Drug: Placebo (PBO)

INTERVENTIONS:
Drug: Vaniprevir — Participants took capsules containing 100 mg Vaniprevir twice daily (b.i.d.), three in the morning (300 mg and 600 mg regimens) and three in the evening (600 mg regimen only), orally, for 24 or 48 weeks.
  Other Names: MK-7009
  Arms: 24-wk Vaniprevir 600 mg + 24-wk PBO + Peg-IFN/RBV; 24-wk Vaniprevir 600 mg + Peg-IFN/RBV; 48-wk Vaniprevir 300 mg + Peg-IFN/RBV; 48-wk Vaniprevir 600 mg + Peg-IFN/RBV
Drug: Pegylated Interferon (Peg-IFN) — Participants used prefilled syringe containing 180 µg/0.5 mL Peg-IFN, for weekly subcutaneous injection, for 24 or 48 weeks
  Other Names: PEGASYS™
Drug: Ribavirin (RBV) — Participants took tablets containing 200 mg RBV, 5 or 6 tablet dosage based on the participant's weight, with food, for 24 or 48 weeks. The dose was 1000 mg for participants weighing <=75 kg and 1200 mg for participants weighing >75 kg.
  Other Names: COPEGUS™
Drug: Placebo (PBO) — Participants took PBO capsules matching Vaniprevir capsules, three in the morning and three in the evening, for 24 or 48 weeks.
  Arms: 24-wk Vaniprevir 600 mg + 24-wk PBO + Peg-IFN/RBV; 48-wk PBO + Peg-IFN/RBV

SUMMARY:
The purpose of this study is to test the safety, tolerability, and efficacy of 4 regimens of Vaniprevir + Peg-IFN and Ribavirin as compared to Placebo (PBO) + Peg-IFN/RBV. The primary hypotheses are that Vaniprevir is well tolerated, and that Vaniprevir 600 mg twice daily (b.i.d.) is superior to the control regimen for the percentage of non-cirrhotic (NC) participants achieving undetectable HCV ribonucleic acid (RNA) 24 weeks after the end of study therapy (SVR24).

ELIGIBILITY:
Inclusion criteria:

* Has chronic HCV genotype 1 infection
* Is treatment-experienced
* For the non-cirrhotic population, has had a liver biopsy without evidence of cirrhosis and hepatocellular carcinoma; for the cirrhotic population, has had a liver biopsy with evidence of cirrhosis and without evidence of hepatocellular carcinoma.

Exclusion criteria:

* Has not tolerated previous course peg-IFN and RBV
* Is unlikely to tolerate at least 24 weeks of continuous therapy with Peg-IFN and RBV
* Is co-infected with Human Immunodeficiency Virus (HIV) and/or hepatitis B
* Consumes excessive amounts of alcohol
* Has a history of drug or alcohol abuse
* If female, participant is pregnant or breastfeeding
* Has been in a clinical trail with an investigational drug in the last 30 days
* Has used IFN/Peg-IFN and RBV in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2009-03-27 (Actual); Primary Completion 2012-03-26 (Actual); Study Completion 2012-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Rodriguez-Torres M, Stoehr A, Gane EJ, Serfaty L, Bhanja S, Barnard RJ, An D, Gress J, Hwang P, Mobashery N. A phase 2B study of MK-7009 (vaniprevir) in patients with genotype 1 HCV infection who have failed previous pegylated interferon and ribavirin treatment. J Hepatol. 2013 Jul;59(1):11-7. doi: 10.1016/j.jhep.2013.02.008. Epub 2013 Feb 21. PMID 23439259
- [Result] Rodriguez-Torres M, Stoehr A, Gane EJ, Serfaty L, Lawitz E, Zhou A, Bourque M, Bhanja S, Strizki J, Barnard RJ, Hwang PM, DiNubile MJ, Mobashery N. Combination of vaniprevir with peginterferon and ribavirin significantly increases the rate of SVR in treatment-experienced patients with chronic HCV genotype 1 infection and cirrhosis. Clin Gastroenterol Hepatol. 2014 Jun;12(6):1029-37.e5. doi: 10.1016/j.cgh.2013.09.067. Epub 2013 Oct 10. PMID 24120953
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-009&kw=7009-009&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-cirrhotic (NC) and cirrhotic (C) participants were screened and enrolled separately in this study. The NC population was used for all safety, tolerability, and efficacy outcome measures. Primary analyses of the outcome measures only included the NC population. Adverse events (AEs) were monitored in both the NC and C populations.
Groups:
- 24-wk Vaniprevir 600 mg + Peg-IFN/RBV: Vaniprevir 600 mg and RBV (1000 mg or 1200 mg total daily dose based on body weight) twice daily (b.i.d.) and peg-IFN 180 mcg injection once weekly for 24 weeks.
- 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV: Vaniprevir 600 mg and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and peg-IFN 180 mcg injection once weekly for 24 weeks, followed by PBO and RBV (1000 mg or 1200 mg based on body weight) b.i.d. and peg-IFN 180 mcg injection once weekly for an additional 24 weeks.
- 48-wk Vaniprevir 300 mg + Peg-IFN/RBV: Vaniprevir 300 mg and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and peg-IFN 180 mcg injection once weekly for 48 weeks.
- 48-wk Vaniprevir 600 mg + Peg-IFN/RBV: Vaniprevir 600 mg and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and peg-IFN 180 mcg injection once weekly for 48 weeks.
- 48-wk PBO + Peg-IFN/RBV: PBO and RBV (1000 mg or 1200 mg total daily dose based on body weight) twice daily (b.i.d.) and Peg-IFN 180 mcg injection once weekly for 48 weeks.
Period: Overall Study (NC Population)
Arm/Group | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Started | 42 | 44 | 41 | 42 | 42
Completed | 37 | 40 | 38 | 38 | 37
Not Completed | 5 | 4 | 3 | 4 | 5
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1
Period: Overall Study (C Population)
Arm/Group | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Started | 16 | 14 | 15 | 15 | 14
Completed | 15 | 11 | 14 | 14 | 14
Not Completed | 1 | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Population consists of all randomized C and NC participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV | Total
Number analyzed (Participants) | 58 | 58 | 56 | 57 | 56 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.0 (8.4) | 51.6 (8.1) | 50.6 (7.5) | 52.1 (8.7) | 49.9 (7.8) | 50.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 16 | 19 | 21 | 105
  Male | 33 | 34 | 40 | 38 | 35 | 180

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SVR24 Following Treatment With Vaniprevir 600 mg b.i.d.
Description: The percentage of non-cirrhotic participants with undetectable Hepatits C virus (HCV) ribonucleic acid (RNA) 24 weeks after completing treatment was determined for each Vaniprevir 600 mg b.i.d. and control regimen. Results for Vaniprevir 300 mg are presented as a Secondary Outcome Measure.
Time Frame: Up to 72 weeks
Population: The Full Analysis Set (FAS) population consists of all non-cirrhotic participants who received at least 1 dose of study treatment, have post-dose endpoint data, and have baseline data for measures that require baseline data.
Measure: Number; unit: Percentage of participants
Groups:
- 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV: Vaniprevir 600 mg and RBV (1000 mg or 1200 mg total daily dose based on body weight) twice daily (b.i.d.) and Peg-IFN 180 mcg injection once weekly for 24 or 48 weeks.
Arm/Group | 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Number analyzed (Participants) | 38 | 38 | 41 | 42
Percentage of participants | 71.1 | 84.2 | 78.0 | 19.0
Statistical Analysis 1: Comparison: 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV vs 48-wk PBO + Peg-IFN/RBV; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in percentage = 53.6, 95% CI 2-sided [34.5 to 69.1] — Adjusted difference subtracts the percentage of PBO-treated participants (i.e., 19.0%) that achieved SVR24 and stratifies by prior treatment response
Statistical Analysis 2: Comparison: 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV vs 48-wk PBO + Peg-IFN/RBV; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in percentage = 64.4, 95% CI 2-sided [45.2 to 78.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 48-wk Vaniprevir 600 mg + Peg-IFN/RBV vs 48-wk PBO + Peg-IFN/RBV; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Adjusted difference in percentage = 59.0, 95% CI 2-sided [40.2 to 73.4] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of non-cirrhotic participants experiencing AEs during the active Vaniprevir/PBO treatment and 14-day follow-up periods was monitored for each treatment regimen. An AE was defined as any unfavorable and unintended change in the structure (signs), function (symptoms), or chemistry (laboratory data) of the body temporally associated with any use of a Sponsor product, whether or not considered related to the use of the product.
Time Frame: Up to 73 weeks
Population: The All-Patients-as-Treated (APaT) population was employed for safety analyses. The APaT population consists of all non-cirrhotic randomized patients who received at least one dose of study treatment.
Measure: Number; unit: Number of participants
Arm/Group | 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Number analyzed (Participants) | 40 | 42 | 41 | 46 | 42
Number of participants | 38 | 42 | 40 | 46 | 41

3. Primary Outcome: Number of Participants Discontinuing From Study Treatment Due to AEs
Description: The number of non-cirrhotic participants withdrawing from study treatment due to AEs during the active Vaniprevir/PBO treatment and 14-day follow-up periods was monitored for each treatment regimen.
Time Frame: Up to 48 weeks
Population: The All-Patients-as-Treated (APaT) population was employed for safety analyses. The APaT population consists of all randomized non-cirrhotic patients who received at least one dose of study treatment.
Measure: Number; unit: Number of participants
Arm/Group | 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Number analyzed (Participants) | 40 | 42 | 41 | 46 | 42
Number of participants | 2 | 3 | 2 | 4 | 1

4. Secondary Outcome: Percentage of Participants Achieving SVR24 Following Treatment With Vaniprevir 300 mg b.i.d.
Description: The percentage of non-cirrhotic participants treated with Vaniprevir 300 mg b.i.d. with undetectable HCV RNA 24 weeks after completing treatment was determined.
Time Frame: 72 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Number analyzed (Participants) | 39 | 42
Percentage of participants | 66.7 | 19.0
Statistical Analysis 1: Comparison: 48-wk Vaniprevir 300 mg + Peg-IFN/RBV vs 48-wk PBO + Peg-IFN/RBV; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen; Adjusted difference in percentage = 47.3, 95% CI 2-sided [29.2 to 63.2] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants Achieving cEVR
Description: The percentage of non-cirrhotic participants with complete early viral response (cEVR; undetectable HCV RNA at Week 12) was determined for each Vaniprevir dose. Since each of the Vaniprevir 600 mg arms had the same treatment history at this point in the study, the data were pooled for analysis.
Time Frame: Up to Week 60
Population: The Full Analysis Set (FAS) population consists of all non-cirrhotic participants who received at least 1 dose of study treatment, have post-dose endpoint data, and have baseline data for measures that require baseline data. The 3 Vaniprevir 600 mg b.i.d. arms were combined in this analysis.
Measure: Number; unit: Percentage of participants
Groups:
- PBO + Peg-IFN/RBV: PBO and RBV (1000 mg or 1200 mg total daily dose based on body weight) b.i.d. and Peg-IFN 180 mcg injection once weekly for 48 weeks.
Arm/Group | 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | PBO + Peg-IFN/RBV
Number analyzed (Participants) | 125 | 41 | 42
Percentage of participants | 92.0 | 85.4 | 9.5
Statistical Analysis 1: Comparison: 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV vs PBO + Peg-IFN/RBV; Test type: Superiority or Other; Adjusted difference in percentage = 82.6, 95% CI 2-sided [69.5 to 90.2] — Adjusted difference subtracts the percentage of PBO-treated participants (i.e., 9.5%) that achieved cEVR and stratifies by prior treatment response
Statistical Analysis 2: Comparison: 48-wk Vaniprevir 300 mg + Peg-IFN/RBV vs PBO + Peg-IFN/RBV; Test type: Superiority or Other; Adjusted difference in percentage = 76.1, 95% CI 2-sided [60.1 to 86.7] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percentage of Participants Achieving SVR24 After 24 Weeks of Vaniprevir 600 mg b.i.d.
Description: The percentage of participants achieving SVR24 after the 24-week Vaniprevir 600 mg b.i.d. regimen at Week 48 was compared to the control regimen.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Number analyzed (Participants) | 38 | 41
Percentage of participants | 71.1 | 36.6
Statistical Analysis 1: Comparison: 24- or 48-wk Vaniprevir 600 mg + Peg-IFN/RBV vs 48-wk PBO + Peg-IFN/RBV; Test type: Superiority or Other; Miettinen and Nurminen method; Adjusted difference in percentage = 35.8, 95% CI 2-sided [15.5 to 53.4] — Adjusted difference subtracts the percentage of PBO patients (36.6%) with undetectable HCV RNA at Week 48 and stratifies by prior treatment response

ADVERSE EVENTS:
Time Frame: AEs were monitored for 50 weeks (48 weeks of active treatment and 2 weeks of follow-up) and serious AEs were monitored for 18 months.
Description: AEs were monitored and presented for the combined NC and C participant populations.
Arm/Group | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV | 48-wk PBO + Peg-IFN/RBV
Serious Adverse Events (participants affected / at risk) | 2/56 | 5/56 | 6/56 | 9/61 | 1/56
Other Adverse Events (participants affected / at risk) | 53/56 | 56/56 | 55/56 | 61/61 | 55/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV (N=56) | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV (N=56) | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV (N=56) | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV (N=61) | 48-wk PBO + Peg-IFN/RBV (N=56)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal vascular thorombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24-wk Vaniprevir 600 mg + Peg-IFN/RBV (N=56) | 24-wk Vaniprevir 600 mg, 24-wk PBO + Peg-IFN/RBV (N=56) | 48-wk Vaniprevir 300 mg + Peg-IFN/RBV (N=56) | 48-wk Vaniprevir 600 mg + Peg-IFN/RBV (N=61) | 48-wk PBO + Peg-IFN/RBV (N=56)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 15 (23) | 12 (16) | 8 (9) | 8 (11)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 1 (6) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (12) | 8 (14) | 8 (25) | 9 (9) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (3) | 3 (3) | 3 (3) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (6) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Conjunctivitis (Eye disorders) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (3) | 5 (5) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 5 (5) | 4 (10) | 8 (8) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 2 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 9 (10) | 5 (6) | 10 (11) | 7 (7)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 23 (40) | 26 (34) | 15 (41) | 33 (48) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 15 (20) | 12 (13) | 12 (14) | 7 (11) | 8 (9)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (9) | 4 (5) | 5 (5) | 5 (5) | 2 (2)
Gingivitis (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (3) | 3 (4) | 2 (2) | 2 (3) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 26 (31) | 25 (27) | 20 (30) | 39 (50) | 10 (10)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 18 (20) | 16 (30) | 8 (11) | 17 (26) | 3 (5)
Asthenia (General disorders) | 12 (12) | 14 (14) | 11 (13) | 13 (14) | 11 (12)
Chest pain (General disorders) | 1 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 4 (4) | 5 (5) | 5 (6) | 2 (2) | 1 (1)
Fatigue (General disorders) | 26 (31) | 22 (26) | 25 (29) | 19 (19) | 18 (20)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 12 (16) | 10 (10) | 17 (18) | 15 (21) | 12 (14)
Injection site erythema (General disorders) | 2 (7) | 3 (3) | 3 (3) | 2 (3) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Irritability (General disorders) | 4 (5) | 6 (6) | 6 (6) | 8 (8) | 8 (8)
Mucosal dryness (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (2) | 2 (4) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 8 (9) | 8 (8) | 9 (12) | 12 (13) | 14 (18)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (3) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 6 (10) | 4 (5) | 4 (4) | 3 (3)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 3 (6) | 4 (6)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6) | 3 (3) | 3 (5) | 5 (5)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (8)
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (3)
Weight decreased (Investigations) | 3 (3) | 0 (0) | 5 (5) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 9 (11) | 14 (15) | 9 (10) | 8 (8) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 8 (8) | 8 (10) | 11 (12) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 6 (6) | 4 (4) | 8 (10) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (3) | 6 (7) | 6 (8) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (8) | 15 (16) | 11 (11) | 12 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 4 (6) | 7 (7) | 5 (5) | 7 (7) | 6 (6)
Dysgeusia (Nervous system disorders) | 5 (5) | 4 (4) | 6 (6) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 23 (36) | 18 (19) | 28 (40) | 23 (34) | 20 (26)
Paraesthesia (Nervous system disorders) | 2 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 5 (6) | 2 (2) | 2 (2) | 3 (3)
Depressed mood (Psychiatric disorders) | 1 (1) | 3 (4) | 7 (9) | 3 (3) | 4 (4)
Depression (Psychiatric disorders) | 4 (4) | 7 (8) | 11 (11) | 10 (10) | 3 (4)
Insomnia (Psychiatric disorders) | 7 (9) | 8 (10) | 17 (18) | 8 (15) | 14 (14)
Mood swings (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 7 (8) | 8 (8) | 7 (7) | 8 (9) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 20 (28) | 9 (10) | 17 (19) | 14 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 9 (9) | 9 (9) | 8 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7) | 1 (1) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 4 (6) | 3 (3) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 4 (4) | 6 (7) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 6 (6) | 9 (9) | 12 (12) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 6 (7) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (12) | 8 (8) | 9 (10) | 10 (10) | 10 (11)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6) | 6 (7) | 7 (7) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (21) | 19 (21) | 17 (23) | 21 (23) | 14 (15)
Rash (Skin and subcutaneous tissue disorders) | 8 (10) | 7 (10) | 8 (9) | 20 (22) | 10 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.